CLINICAL TRIAL: NCT03668184
Title: What Are the Predictive Factors for Preeclampsia in Oocyte Recipients? - PREROVE
Acronym: PREROVE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3078_PREROVE
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy; Oocyte Donation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: preeclampsia — occurrence of pre-eclampsia

SUMMARY:
The main goal is to determine which risk factors develop preeclampsia in this specific group of oocyte recipients.

ELIGIBILITY:
Inclusion Criteria:

* All major patients with a pregnancy of more than 22 weeks of amenorrhea resulting from an oocyte donation in one of the study centers, having given birth between January 2010 and April 2017 and not opposed to participation in the study.

Exclusion Criteria:

* all pregnancies resulting from an oocyte donation abroad, persons of legal age subject to legal protection (safeguard of justice, guardianship, tutorship) and persons deprived of their liberty.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with a pregnancy of more than 22 weeks of amenorrhea resulting from an oocyte donation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
occurrence of pre-eclampsia | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Solène DUROS, MD, Principal Investigator — Rennes University Hospital
Locations (2):
- France (2):
  - CHU de Rennes, Rennes
  - Clinique de la sagesse, Rennes